CLINICAL TRIAL: NCT04404842
Title: Development of a Screening Tool for the Risk of Vitamin D Deficiency
Acronym: EvidenceQ
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Pavia (Other)
Collaborators: Istituti Clinici Scientifici Maugeri SpA (Other)
Responsible Party: Principal Investigator, Hellas Cena, Tenured researcher, University of Pavia
Other Study IDs: 14052020
Record Dates: First submitted 2020-05-18; First posted 2020-05-28 (Actual); Last update posted 2020-05-28 (Actual); Status verified 2020-05

CONDITIONS: Vitamin D Deficiency; Vitamin D3 Deficiency; Vitamin D
Keywords: Vitamin D; Cholecalciferol; Deficiency; Inadeguacy; Screening; Questionnaire; Survey
MeSH Terms: conditions — Vitamin D Deficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- EvidenceQ Cohort: Adult subjects, aged over 18 years, male and female.

SUMMARY:
Since vitamin D deficiency is a condition that affects a high percentage of individuals of all ages and given the attention on the possible role of the deficiency of this vitamin in the development of various chronic diseases, including cardiovascular and metabolic disease (obesity, insulin resistance, hypertension, diabetes) and the correlation with mortality from major cardiovascular events (heart failure, myocardial infarction, sudden cardiac death, stroke, atrial fibrillation and peripheral vascular disease), it is clear that in clinical practice it is necessary to provide screening tools characterized by a simple use, high efficacy and a low economic impact, useful to detect a possible deficiency state that has a significant impact on general health and therefore provide targeted interventions for diagnosis and supplementation when and if necessary. Therefore, the objective of this study project is part of the broader context of supporting, with reproducible and shared scientific data, operational protocols useful for the clinician to identify subjects potentially at risk of vitamin D deficiency as well as directing to the diagnostic and more effective therapeutic. Surveillance of vitamin D status should be a high priority in which easy-to-use and interpreted tools, such as the questionnaire developed for this study, could respond to the needs of early identification of subjects potentially at risk of hypovitaminosis D, thus supporting the work of the clinician.

DETAILED DESCRIPTION:
It will be administered the questionnaire which includes specific and previously identified questions useful for the purpose of the study to all patients who belong to the clinic of the Dietetics and Clinical Nutrition, Internal Medicine and Endocrinology Unit, ICS Maugeri di Pavia who meet the inclusion criteria and signed the Informed Consent. The blood dosage of 25 (OH) D will be used as a reference standard useful for achieving the purpose of the study subject to the execution of diagnostic-therapeutic procedures that are beneficial to the patient or performed for routine diagnostic procedures or previously prescribed by the general practitioner. The collected data will be entered in the Data Collected Form together with the laboratory tests.

Therefore, all patients will receive the EVIDENCE Questionnaire which includes 19 items that investigate those factors that influence the production, absorption and intake of vitamin D:

* anthropometric data (weight, height, waist circumference, BMI),
* demographic information, such as latitude and phototype,
* dietary intake of vitamin D,
* health status and therapies,
* multivitamin or vitamin D supplementation,
* sun exposure habits according to the season, frequency and time of exposure, the body parts exposed, the sunscreens use and outdoor activities.

The aim of the study is to develop a questionnaire useful in screening the adequacy of vitamin D concentration in the adult population and to produce evidence of construct validity and concurrent validity of the questionnaire itself.

SAMPLE SIZE: Psychometric literature suggests enrolling around 5-10 subjects for each item. Considering the number of items in the questionnaire, equal to 19, the number of subjects to be enrolled will be approximately 190.

ELIGIBILITY:
Inclusion Criteria:

* Subjects older than or equal 18 years;
* Absence of liver pathologies;
* Absence of kidney pathologies;
* Absence of intestinal malabsorption syndromes;
* Absence of bariatric surgery;
* Absence of cancer;
* Absence of primary hyperparathyroidism;
* Absence of extensive dermatological pathologies (e.g. psoriasis, atopic dermatitis, vitiligo)
* Absence of supplementation with multivitamin supplements or vitamin D;
* Absence of chronic drug therapy with: anticonvulsants, antipsychotics, glucocorticoids, immunosuppressive corticosteroids, anti-retrovirals, slimming, hypocolestrolemicants, laxatives (prolonged use);
* acceptance and sign of informed consent.

Exclusion Criteria:

* Subjects under 18 years old;
* Affected by liver pathologies;
* Affected by kidney pathologies;
* Affected by intestinal malabsorption syndromes;
* Affected by cancer;
* Affected by primary hyperparathyroidism;
* Affected by extensive dermatological pathologies (e.g. psoriasis, atopic dermatitis, vitiligo).
* Candidates and/or undergoing bariatric surgery;
* Supplementation with multivitamin or vitamin D;
* Chronic therapy with: anticonvulsants, antipsychotics, glucocorticoids, immunosuppressive corticosteroids, anti-retrovirals, slimming, hypocolestrolemizzanti, laxatives (prolonged use).

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Psychometric literature suggests that about 5-10 subjects should be recruited for each item (Steiner DL et al, 2015). Considering the number of items in the questionnaire, equal to 19, the number of subjects to enlist will be about 190.
  Consecutively recruited adult patients by the Service of Dietetics and Clinical Nutrition, Unit of Internal Medicine and Endocrinology, of both sexes.
Sampling Method: Probability Sample
Enrollment: 190 (Estimated)
Dates: Start 2020-01-14 (Actual); Primary Completion 2022-01-31 (Estimated); Study Completion 2022-01-31 (Estimated)

PRIMARY OUTCOMES:
Construct validity (EVIDENCE Questionnaire) | 1 hour
  The construct validity of the questionnaire will be assessed using exploratory factorial analysis.
Internal consistency (EVIDENCE Questionnaire) | 1 hour
  The internal consistency will be evaluated with the Cronbach alpha coefficient or with the McDonald Omega coefficient.
Concurrent validity (EVIDENCE Questionnaire) | 1 hour
  The concurrent validity will be assessed by comparing the results obtained with the serum 25 (OH) D dosage taken as the reference standard.
Questionnaire Scoring | 1 hour
  Determine the optimal cut-off score of EvidenceQ for screening of subjects potentially at risk of vitamin D inadequacy.

CONTACTS AND LOCATIONS:
Overall Officials: Hellas Cena, Principal Investigator — Univeristy of Pavia, ICS Maugeri SpA SB
Locations (1):
- Istituti Clinici Scientifici Maugeri SpA, Pavia, Lombardy, Italy